CLINICAL TRIAL: NCT07208734
Title: Development and Multicenter Validation of a Personalized Transcranial Alternating Current Stimulation Protocol for Cognitive Impairment in Older Adults
Brief Title: Personalized Brain Stimulation for Cognitive Impairment in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025116
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer s Disease
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Alternating Current Stimulation (tACS) or AI-based Cognitive Training (Experimental)
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS); Other: AI-based Cognitive Training
- Sham intervention (Sham Comparator)
  Interventions: Other: Sham intervention

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation (tACS) — Gamma TranscraniaThis intervention uses a personalized transcranial alternating current stimulation (tACS) protocol specifically designed for older adults with cognitive impairment. Unlike standard brain stimulation approaches, this protocol is individualized through artificial intelligence-based modeling of each participant's brain imaging data to optimize electric field distribution. The study will evaluate both safety and effectiveness in a multicenter randomized controlled trial.l Alternating Current Stimulation (tACS)
  Arms: Transcranial Alternating Current Stimulation (tACS) or AI-based Cognitive Training
Other: AI-based Cognitive Training — This intervention provides a personalized cognitive training program tailored to multiple cognitive domains. Using algorithm-based task matching, the system delivers training exercises adapted to each participant's cognitive profile. The program is designed to target memory, attention, executive function, and language, and will be validated through a multicenter randomized controlled trial.
  Arms: Transcranial Alternating Current Stimulation (tACS) or AI-based Cognitive Training
Other: Sham intervention — The sham stimulation group will undergo the same setup procedures as the active tACS group, including electrode placement and device operation. However, no effective current will be delivered beyond an initial brief sensation, ensuring participants cannot distinguish sham from active stimulation. This allows blinding of participants and investigators to treatment allocation.
  Arms: Sham intervention

SUMMARY:
This study aims to develop and test new personalized treatments for older adults with cognitive impairment.

Project 1: Create a personalized cognitive training program using computer algorithms to match training tasks to individual needs. About 300 participants will join a randomized trial at hospitals and community health centers.

Project 2: Develop a personalized brain stimulation program (tACS) based on brain imaging and artificial intelligence. About 160 participants will be enrolled to test safety and effectiveness.

Project 3: Build a framework for ethical data management by reviewing international practices and consulting experts.

Together, these projects will provide evidence for safe, effective, and personalized care, while ensuring responsible use of research data.

DETAILED DESCRIPTION:
This study is designed to improve the treatment and care of older adults with cognitive impairment through three related projects.

Project 1: Development of a personalized cognitive training program. Using advanced computer algorithms, we will match training tasks to each patient's needs across multiple cognitive domains. About 300 participants will be enrolled from hospitals and community health centers in two provinces to test the effectiveness of this program in a randomized controlled trial.

Project 2: Development of a personalized brain stimulation program. Based on brain imaging data and artificial intelligence models, we will create individualized transcranial alternating current stimulation (tACS) plans to deliver precise, safe, and effective stimulation. About 160 participants will be recruited from the same sites to evaluate safety and effectiveness in a randomized controlled trial.

Project 3: Development of a data governance and ethics framework. Building on the first two projects, we will review international literature and consult experts in ethics, geriatrics, neuroscience, and data governance to create a framework for managing multimodal data and ethical issues in cognitive impairment research.

Together, these projects aim to provide personalized, scientifically validated treatment strategies and ensure that research data are managed safely and ethically.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients or outpatients aged 50-90 years;
2. Patients diagnosed with amnestic mild cognitive impairment (aMCI) due to AD or mild dementia due to AD, based on the 2018 NIA-AA clinical diagnostic criteria established by the National Institute on Aging and the Alzheimer's Association;
3. Neuropsychological assessment showing MMSE scores between 18 and 26, and a CDR score of 0.5 or 1;
4. Able to communicate fluently in Chinese (non-illiterate);
5. For those currently receiving cholinesterase inhibitor therapy (e.g., donepezil or rivastigmine), the treatment dose must be stable, defined as a fixed dosage administered continuously for at least six weeks, with no adjustment of the medication regimen during the study period;
6. Provision of written informed consent.

Exclusion Criteria:

1. Documented history of cerebrovascular stroke, with clear neurological deficits at onset and corresponding responsible lesions on neuroimaging;
2. Moderate to severe white matter lesions (Fazekas score 3-6);
3. Presence of any cause of consciousness disorder;
4. Severe aphasia or motor disability that prevents completion of neuropsychological assessments;
5. Current psychiatric disorders;
6. History of alcohol dependence, drug addiction, traumatic brain injury, epilepsy, encephalitis, normal-pressure hydrocephalus, or other neurological disorders that may cause cognitive impairment;
7. Systemic diseases that may contribute to mild cognitive impairment (e.g., hepatic or renal insufficiency, endocrine disorders, vitamin deficiencies);
8. Considered unsuitable for participation by the investigators.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Moca score | Participants will undergo a screening period, a baseline period, an 8-week visit, and a 6-month visit (calculated from the first intervention) during the trial.

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-cog, 11-items version). | Participants will undergo a screening period, a baseline period, an 8-week visit, and a 6-month visit (calculated from the first intervention) during the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing 100053, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided